CLINICAL TRIAL: NCT06173869
Title: A Randomised, Controlled, Assessor-blind, Parallel Groups, Multicentre Trial Comparing the Ovarian Response of a Starting Dose of Either 10 μg or 15 μg Follitropin Delta (FE 999049) to a Starting Dose of Either 150 IU or 225 IU Follitropin Alfa (GONAL-F) in Conventional Regimens in Controlled Ovarian Stimulation in Women Undergoing an Assisted Reproductive Technology Programme in China
Brief Title: A Randomised Trial Comparing the Ovarian Response of a Starting Dose of Either 10 μg or 15 μg Follitropin Delta (FE 999049) to a Starting Dose of Either 150 IU or 225 IU Follitropin Alfa (GONAL-F) in Conventional Regimens in China
Acronym: COCO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 000413
Record Dates: First submitted 2023-12-06; First posted 2023-12-18 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — FE 999049; follitropin delta; follitropin alfa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FE 999049 (Experimental): The participants receive either low or high starting dose as appropriate according to Investigators Judgement.
  10 or 15 µg
  Interventions: Drug: FE 999049
- GONAL-F (Active Comparator): The participants receive either low or high starting dose as appropriate according to Investigators Judgement.
  150 or 225 IU.
  Interventions: Drug: GONAL-F

INTERVENTIONS:
Drug: FE 999049 — FE 999049 was administered as single daily subcutaneous injections at a starting dose of either 10 or 15 µg daily that was fixed for the first five stimulation days. Based on ovarian response, the dose could be increased or decreased by 5 µg, with dose adjustments implemented not more frequently than once every 2 days per investigator's judgement. The minimum daily dose was 5 µg, and the maximum daily dose was 20 µg. Participants could be treated for a maximum of 20 days.
  Other Names: Rekovelle; Follitropin Delta
  Arms: FE 999049
Drug: GONAL-F — GONAL-F was administered as single daily subcutaneous injections at a starting dose of either 150 or 225 IU daily that was fixed for the first five stimulation days. Based on ovarian response, the dose could be increased or decreased by 75 IU, with dose adjustments implemented not more frequently than once every 2 days per investigator's judgement. The minimum daily dose was 75 IU, and the maximum daily dose was 300 IU. Participants could be treated for a maximum of 20 days.
  Coasting was not allowed.
  Arms: GONAL-F

SUMMARY:
This is a phase 3b clinical trial with follitropin delta (FE 999049) and Gonal-F. The trial is a randomised, controlled, assessor-blind, parallel groups, multicentre trial comparing the ovarian response of a starting dose of either 10mg or 15 mg follitropin delta to a starting dose of either 150 IU or 225 IU Gonal-F in a long GnRH agonist protocol in women undergoing an assisted reproductive technology programme in China.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated Informed Consent Form for participation in the trial, obtained before any trial-related procedures.
* In good physical and mental health in the judgement of the investigator.
* Chinese pre-menopausal female between the ages of 20 and 40 years; at least 20 years (including the 20th birthday) when signing the informed consent and no more than 40 years (up to the day before the 41st birthday) at the time of randomisation.
* Eligible for ovarian stimulation with a dose equivalent to 150 IU GONAL-F or 225 IU GONAL-F, as judged by the investigator.
* Body mass index (BMI) between 17.5 and 32.0 kg/m2 (both inclusive) at screening.
* Infertile women diagnosed with tubal infertility, unexplained infertility, endometriosis stage I/II or with partners diagnosed with male factor infertility, eligible for in vitro fertilisation (IVF) or intracytoplasmic sperm injection (ICSI) using fresh or frozen ejaculated sperm from male partner or sperm donor
* Infertility for at least one year before randomisation for subjects <35 years or for at least 6 months for subjects ≥35 years (criteria not applicable in case of tubal or severe male factor infertility).
* Regular menstrual cycles of 24-35 days (both inclusive), presumed to be ovulatory.
* Transvaginal ultrasound documenting presence and adequate visualisation of both ovaries, without evidence of significant abnormality. Both ovaries must be accessible for oocyte retrieval.
* Early follicular phase (cycle day 2-4) serum levels of follicle-stimulating hormone (FSH) between 1 and 15 IU/L (results obtained within 3 months prior to randomisation).
* Serum anti-Müllerian hormone (AMH) concentration of ≤35 pmol/L at screening.

Exclusion Criteria:

* Primary ovarian failure.
* More than three previous controlled ovarian stimulation cycles initiated, regardless of outcome.
* History of previous episode of OHSS, exuberant ovarian response to gonadotropins, or polycystic ovarian syndrome.
* Known endocrine or metabolic abnormalities (pituitary, adrenal, pancreas, liver or kidney) which can compromise participation in the trial with the exception of controlled thyroid function disease.
* Known tumours of the ovary, breast, uterus, adrenal gland, pituitary or hypothalamus which would contraindicate the use of gonadotropins.
* Fibroid tumours of the uterus incompatible with pregnancy.
* Currently breast-feeding.
* Known inherited or acquired thrombophilia disease.
* Active arterial or venous thromboembolism or severe thrombophlebitis, or a history of these events.
* Known porphyria.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 301 (Actual)
Dates: Start 2024-03-29 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (11):
- China (11):
  - Ferring Investigational Site, Shushan, Anhui
  - Ferring Investigational Site, Yuzhong, Chongqing Municipality
  - Ferring Investigational Site, Guangzhou, Guandong
  - Ferring Investigational Site, Guangzhou, Guangdong
  - Ferring Investigational Site, Zhengzhou, Henan
  - Ferring Investigational Site, Nanchang, Jiangxi
  - Ferring Investigational Site, Shengyang, Liaoling
  - Ferring Investigational Site, Shanghai, Shanghai Municipality
  - Ferring Investigational Site, Chengdu, Sichuang
  - Ferring Investigational Site, Tianjin, Tianjin Municipality
  - Ferring Investigational Site, Xiaobailou, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- FE 999049: The participants received either low or high starting dose as appropriate according to Investigators Judgement.
  10 or 15 µg
  FE 999049: FE 999049 was administered as single daily subcutaneous injections at a starting dose of either 10 or 15 µg daily that was fixed for the first five stimulation days. Based on ovarian response, the dose was increased or decreased by 5 µg, with dose adjustments implemented not more frequently than once every 2 days per investigator's judgement. The minimum daily dose was 5 µg, and the maximum daily dose was 20 µg. Participants were treated for a maximum of 20 days.
- GONAL-F: The participants received either low or high starting dose as appropriate according to Investigators Judgement.
  150 or 225 IU.
  GONAL-F: GONAL-F was administered as single daily subcutaneous injections at a starting dose of either 150 or 225 IU daily that was fixed for the first five stimulation days. Based on ovarian response, the dose was increased or decreased by 75 IU, with dose adjustments implemented not more frequently than once every 2 days per investigator's judgement. The minimum daily dose was 75 IU, and the maximum daily dose was 300 IU. Participants were treated for a maximum of 20 days.
  Coasting was not allowed.
Period: Overall Study
Arm/Group | FE 999049 | GONAL-F
Started | 148 | 153
Completed | 126 | 131
Not Completed | 22 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FE 999049 | GONAL-F | Total
Number analyzed (Participants) | 148 | 153 | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (3.6) | 32.2 (3.8) | 32.3 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 153 | 301
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 148 | 153 | 301
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 148 | 153 | 301
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 148 | 153 | 301
Dose Group [Count of Participants; unit: Participants]
  Low Starting Dose | 47 | 51 | 98
  High Starting Dose | 101 | 102 | 203
Body Measurement (Weight) [Mean (Standard Deviation); unit: kg] | 57.5 (8.3) | 57.5 (7.7) | 57.5 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Oocytes Retrieved
Time Frame: On day of oocyte retrieval (up to 22 days after start of stimulation)
Measure: Mean (Standard Deviation); unit: Oocytes retrieved
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Oocytes retrieved | 12.7 (5.2) | 11.8 (5.3)

2. Secondary Outcome: Number of Follicles on Stimulation Day 6 and End-of-stimulation
Time Frame: Stimulation day 6 and end-of-stimulation (maximum stimulation day 20)
Measure: Mean (Standard Deviation); unit: Follicles
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Follicles
  Stimulation day 6 | 2.9 (3.0) | 3.0 (3.3)
  End of stimulation | 13.3 (4.4) | 12.7 (4.5)

3. Secondary Outcome: Serum Concentrations of Estradiol on Stimulation Day 6 and End-of-stimulation
Time Frame: stimulation day 6 and end-of-stimulation (maximum stimulation day 20)
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 147 | 153
pmol/L
  Stimulation day 6 | 1303.2 (1093.1) | 1275.9 (1050.8)
  End of stimulation | 11181.2 (5842.2) | 10124.1 (4522.2)

4. Secondary Outcome: Serum Concentrations of Progesterone on Stimulation Day 6 and End-of-stimulation
Time Frame: stimulation day 6 and end-of-stimulation (maximum stimulation day 20)
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
nmol/L
  Stimulation day 6 | 1.6 (0.9) | 1.4 (0.8)
  End of Stimulation | 3.4 (1.6) | 2.8 (1.3)

5. Secondary Outcome: Number of Fertilised Oocytes
Time Frame: On day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Measure: Mean (Standard Deviation); unit: Fertilised Oocytes
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Fertilised Oocytes | 7.8 (4.3) | 7.4 (4.3)

6. Secondary Outcome: Fertilisation Rate
Time Frame: On day 1 after oocyte retrieval (up to 23 days after start of stimulation)
Measure: Mean (Standard Deviation); unit: percentage of fertilised oocytes
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 151
percentage of fertilised oocytes | 59.6 (19.9) | 62.7 (20.9)

7. Secondary Outcome: Number of Embryos (Total and Quality)
Time Frame: Day 3 after oocyte retrieval
Measure: Mean (Standard Deviation); unit: Embryos
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Embryos
  Total | 8.8 (4.6) | 8.2 (4.6)
  Good-Quality | 5.5 (3.7) | 5.1 (3.7)

8. Secondary Outcome: Total Gonadotropin Dose
Time Frame: Up to 20 stimulation days
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
ug | 154.1 (41.0) | 167.7 (48.4)

9. Secondary Outcome: Number of Stimulation Days
Time Frame: Up to 20 stimulation days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
days | 10.6 (1.5) | 10.5 (1.7)

10. Secondary Outcome: Positive βhCG (Positive Serum βhCG Test 13-15 Days After Transfer) Rate
Time Frame: 13-15 days after transfer
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Participants
  Positive | 71 | 72
  Negative | 77 | 81

11. Secondary Outcome: Clinical Pregnancy (at Least One Gestational Sac 5-6 Weeks After Transfer) Rate
Time Frame: 5-6 weeks after transfer
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Participants
  Positive | 61 | 56
  Negative | 87 | 97

12. Secondary Outcome: Vital Pregnancy (at Least One Intrauterine Gestational Sac With Fetal Heart Beat 5-6 Weeks After Transfer) Rate
Time Frame: 5-6 weeks after transfer
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Participants
  Positive | 59 | 50
  Negative | 89 | 103

13. Secondary Outcome: Implantation Rate
Description: The implantation rate was defined as the number of gestational sacs 5-6 weeks after transfer divided by number of embryos transferred.
Time Frame: 5-6 weeks after transfer
Population: Total Number of gestational sacs (subject level)
Measure: Number; unit: percentage of embryos transferred
Units Other Than Participants: Number of transferred embryos
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Number analyzed (Number of transferred embryos) | 185 | 191
percentage of embryos transferred | 40.5 | 62

14. Secondary Outcome: Ongoing Pregnancy (at Least One Intrauterine Viable Fetus 10-11 Weeks After Transfer) Rate
Time Frame: 10-11 weeks after transfer
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Participants
  Positive | 54 | 45
  Negative | 94 | 108

15. Secondary Outcome: Ongoing Implantation Rate (Number of Intrauterine Viable Fetuses 10-11 Weeks After Transfer Divided by Number of Embryos Transferred)
Description: The ongoing implantation rate was defined as the number of intrauterine viable fetuses 10-11 weeks after transfer divided by the number of embryos transferred.
Time Frame: 10-11 weeks after transfer
Population: Low starting dose: 10 μg FE 999049 or 150 IU GONAL-F, high starting dose: 15 μg FE 999049 or 225 IU GONAL-F
Measure: Number; unit: percentage of embryos transferred
Units Other Than Participants: Number of transferred embryos
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Number analyzed (Number of transferred embryos) | 185 | 191
percentage of embryos transferred | 36.2 | 26.2

16. Secondary Outcome: Early Ovarian Hyperstimulation Syndrome (OHSS), Late OHSS, and Total OHSS (All Overall and by Grade)
Description: Early OHSS was defined as OHSS with onset ≤9 days after triggering of final follicular maturation. Late OHSS was defined as OHSS with onset >9 days after triggering of final follicular maturation. Total OHSS measure the incidence of OHSS both early and late.
Time Frame: ≤9 days after triggering of final follicular maturation (early OHSS), >9 days after triggering of final follicular maturation until 21-28 days after last IMP dose or up to ongoing pregnancy 8-9 weeks after transfer in pregnant participants (late OHSS)
Measure: Count of Participants; unit: Participants
Arm/Group | FE 999049 | GONAL-F
Number analyzed (Participants) | 148 | 153
Participants
  Early OHSS | 4 | 8
  Late OHSS | 2 | 1
  Total OHSS | 6 | 9

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | FE 999049 | GONAL-F
All-Cause Mortality (participants affected / at risk) | 0/148 | 0/153
Serious Adverse Events (participants affected / at risk) | 4/148 | 11/153
Other Adverse Events (participants affected / at risk) | 16/148 | 25/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (N=148) | GONAL-F (N=153)
Bartholin's abscess (Infections and infestations) | 0 (0) | 1 (1)
Dengue Fever (Infections and infestations) | 1 (1) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4)
Abortion Threatened (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3)
Ovarian Hyperstimulation Syndrome (Reproductive system and breast disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FE 999049 (N=148) | GONAL-F (N=153)
Upper respiratory tract infection (Infections and infestations) | 9 (10) | 5 (5)
Biochemical Pregnancy (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 15 (15)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 5 (5)
Morning Sickness (Pregnancy, puerperium and perinatal conditions) | 12 (18) | 10 (15)
Hydrometra (Reproductive system and breast disorders) | 9 (9) | 7 (8)
Pelvic discomfort (Reproductive system and breast disorders) | 8 (8) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT06173869/Prot_SAP_000.pdf